CLINICAL TRIAL: NCT01730287
Title: Effect Of Different Lining Materials on Clinical Symptoms of Stepwise Excavation Without Re-enter: Double Blind Randomizd Clinical Trial
Brief Title: Effect Of Different Lining Materials in Stepwise Excavation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sepideh Banava.DDS,MS, Assist-Prof, Azad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AZadUMS-
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Dental Pulp Necrosis
Keywords: Stepwise Excavation; Pulpal vitality; Deep caries lesions; Clinical symptoms; Radiographic evaluation
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Calcium Hydroxide; Dycal; CMW cement; mineral trioxide aggregate; Pemetrexed; calcium-enriched mixture cement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (Experimental): No lining applied in group1.
  Interventions: Drug: Control
- CEM cement (Experimental): CEM cement applied over remained caries in group4.
  Interventions: Drug: CEM cement
- Mineral Trioxide Aggregate (MTA) (Experimental): MTA applied over remained caries in group3.
  Interventions: Drug: Mineral Trioxide Aggregate(MTA)
- Calcium Hydroxide (Experimental): Calcium Hydroxide applied over remained caries in group2.
  Interventions: Drug: Calcium Hydroxide

INTERVENTIONS:
Drug: Control — The teeth in this group restored only by filling material,without liner application.
  Other Names: NO liner applied.
  Arms: Control
Drug: Calcium Hydroxide — Calcium Hydroxide paste applied.
  Other Names: Calcium Hydroxide paste , Dycal,Dentsply.
  Arms: Calcium Hydroxide
Drug: Mineral Trioxide Aggregate(MTA) — MTA applied .
  Other Names: MTA, white MTA, ProRoot,Dentsply.
  Arms: Mineral Trioxide Aggregate (MTA)
Drug: CEM cement — CEM cement applied .
  Other Names: CEM cement, Yektazist,Iran.
  Arms: CEM cement

SUMMARY:
Deep carious lesions will encounter the dentist with the challenge of selecting a treatment method that could avoid the pulpal exposure and maintain the pulp vitality.Conventional restorative treatments suggest complete removal of the caries in one visit which could cause pulpal exposure in 53% of the cases which in next step needs pulpotomy, pulpectomy or Root Canal Therapy (RCT).

Stepwise Excavation(SE)is an old concept but has been researched recently to reduce the possibility pulpal exposure during the removal of the lesion. Contrary to Indirect Pulp Capping (IPC), in this technique only the central infected part of the caries is removed in first visit and the rest of the caries will be lined by a suitable material to suppress the remained cariogenic biomass and seal the cavity. This will help the pulp to defend and survive. After a period, the cavity is re-opened and the rest of the caries which is darker, harder and with less bacteria will be removed and the tooth is restored permanently.The aim of this study was to compare the effect of different lining materials in clinical and radiographical symptoms in stepwise excavation without re-enter after one year.

DETAILED DESCRIPTION:
In this randomized clinical trial of 4 lining materials have been applied in deep caries teeth in stepwise excavation. The common material which is applied as a liner over the remained caries in SE is Calcium Hydroxide(CH). There are several reports of the solubility of this liner over time which could interact with sealing of the cavity in long term. It seems that a material with antibacterial activity, good sealing ability and suitable mechanical properties could cause SE be done efficiently with good prognosis.

MTA is a biomaterial that has been introduced since 1993 with antibacterial property and good sealing ability. A New Endodontic Cement, Calcium Enriched Mixture (CEM) cement with good antibacterial effect like CH with sealing ability that is proposed to be similar to MTA according to its double sealing property. CEM cement has been suggested as a suitable material in pulp capping of permanent molars with irreversible pulpitis.

ELIGIBILITY:
Inclusion Criteria:

A tooth with deep caries lesion - Tooth at risk of pulpal exposure - No pulpal , instantaneous , night pain

Exclusion Criteria:

Unbearable pain of the involved tooth- Apical radiolucency of the tooth- PDL widening

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-12 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Pulpal Vitality | One year
  Clinical symptoms, radiographic evaluation. Sensitivity to cold, hot, pressure, percussion.

CONTACTS AND LOCATIONS:
Overall Officials: Sepideh Banava, Assist-Prof, Study Chair — Azad University of Medical Sciences, Dental Branch - Endodontics research center , SBMU
Locations (1):
- Azad University of Medical Sciences, Dental Branch, Tehran, N/A = Not Applicable, Iran